CLINICAL TRIAL: NCT06196645
Title: Development Of A Physical Activity İntervention Plan Based On The Theory Of Planned Behavior For High School Adolescent Girls
Brief Title: Development of a Planned Behavior Theory-Based Physical Activity Application for High School Adolescent Girls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Technical University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Gunay yildizer, Associate Professor, Eskisehir Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EskisehirTU-SBF-GY02
Record Dates: First submitted 2023-12-26; First posted 2024-01-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Sedentary Lifestyle; Sedentary Behavior; Physical Activity Level
Keywords: Theory of planned behavior; physical activity intervention; adolescent girls
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group-1 (Experimental): Participants in this arm of the experimental group will participate in a school-based intervention program that is based on the theory of planned behavior and includes behavior change techniques. These participants will participate in the intervention plan only in physical education and sports classes at their schools.
  Interventions: Behavioral: Physical Activity Intervention Based on Theory of Planned Behavior
- Control Group (No Intervention): This group will not be involved in any implementation until the end of the research. Ethically, after the research is completed, the proposal to repeat the most effective intervention arm for this group will be presented to the participants in this group.

INTERVENTIONS:
Behavioral: Physical Activity Intervention Based on Theory of Planned Behavior — The content of the intervention plan to be implemented consists of the following components: (I) transferring knowledge about health-related physical fitness and physical activity, (II) taking individual responsibility for physical activity monitoring and simple individual planning, (III) including in the program the types of activities that female adolescents choose and declare that they would enjoy participating in.
  Arms: Intervention Group-1

SUMMARY:
The aim of this study is to examine the effects of a physical activity intervention plan developed based on the theory of planned behavior on the physical activity levels of adolescent girls, their sedentary time and their knowledge about physical activity.

Within the scope of this research, answers to the following research questions will be sought;

1. Is there a difference in physical activity level between participants in the physical activity intervention plan groups and the control group?
2. Is there a difference in terms of daily sedentary time between participants in the physical activity intervention plan groups and the control group?
3. Is there a difference in beliefs about physical activity between participants in the physical activity intervention plan groups and the control group?

In this context, researchers will compare 3 groups within the scope of the data provided by two preliminary studies conducted previously. These groups; (1) intervention group based on the theory of planned behavior, (2) intervention group based on the theory of planned behavior with family participation, (3) control group.

DETAILED DESCRIPTION:
While the physical activity participation of adolescents in Turkey and around the world is quite low, this is more pronounced for girls. The low physical activity participation rates seen in this group shed light on the negative situations to be seen in the future in terms of public health and the economy. The fact that health-related behavior patterns acquired during adolescence form a highly effective basis for the rest of life makes it necessary to develop effective, low-cost physical activity intervention plans for adolescents that take into account individual needs. Research on physical activity intervention, while generally targeting groups with low physical activity levels, is applied in different contexts (school, family, school and family, living environment) where these groups spend their time. In this respect, school-based interventions, where adolescents spend most of their time, come to the fore. For plans to be effective, they should be based on a research process and their theoretical foundations should be inclusive. While the theory of planned behavior, which has an important place in shaping health behaviors and explains the formation and continuity of behavior by addressing the attitude, norms created by the social environment, and the control perceived by the person towards the behavior, constitutes the theoretical basis of this research, the aim of the research is to create and test a school-based physical activity intervention plan based on the theory of planned behavior, targeting adolescent girls.

Qualitative and quantitative research methods were applied through a multi-stage design process, and the findings revealed the need to create an effective intervention plan guide for adolescent girls in Turkish society. These phases included (I) a study to explain which factors are important for physical activity behavior in adolescent girls, including open-ended questions and semi-structured interviews; (II) the process of developing a measurement tool in the light of the data obtained with these qualitative methods; and (III) survey research that adopted the general survey model and reached a large population. As a result of this process, which has been going on for about 48 months, the physical activity intervention plan to be implemented has been shaped. With this intervention, it is aimed to create significant effects among adolescent girls in terms of physical activity and sedentary time and to positively affect their beliefs about physical activity.

The physical activity intervention plan to be developed according to the planned behavior theory will be based on the information obtained in pilot studies that have already been completed. The plan will be implemented in selected high schools affiliated with the Turkish Ministry of National Education. The developed protocol is planned to be implemented over two different time periods. The reason for this is that seasonal factors are emphasized as an important factor in carrying the gains provided in physical activity intervention plans into daily life (Rowland et al., 2006; Tucker & Gililand, 2007; Belanger et al., 2009; Kornides et al., 2018). The contents of the intervention plan will be delivered to students for 2 hours in selected physical education and sports classes. It is planned to implement this plan in physical education classes for one semester. Considering that the implementation will take place in one academic year, data will be collected at the beginning and end of the first semester and at the end of the second semester. Data collection processes are planned to take approximately 1-1.5 months. Thus, it will be ensured that this application will be carried out for 3-3.5 months in a semester. While planning this period, Owen et al. (2017) reviews and meta-analyses were taken into consideration.

Structurally, the physical activity intervention plan is planned to include four dimensions based on the theory of planned behavior. The first two of these are: (I) transferring information on health-related physical fitness and physical activity; (II) taking individual responsibility for physical activity follow-up; and (II) simple individual planning, which will affect the level of physical activity at the individual level. Another dimension is the inclusion in the program of the types of activities that the female adolescents (III) chose and declared that they would enjoy participating in. The last dimension, as emphasized in the theory of planned behavior, is the invitation of significant others, which are the family, teachers, and other students, including male students, with whom the target group is in constant social interaction, to this plan, and all of the practices are open to them. However, data will not collected from them.

ELIGIBILITY:
Inclusion Criteria:

* Bein high school student
* Do not have any health problems that would prevent from participating in exercise,
* Not participating any another exercise/training program during the research process,
* Voluntarily participation -Being suitable for exercise participation according to Physical Activity -- Readiness Questionnaire (PARQ) test results

Exclusion Criteria:

* Presence of any significant health conditions that may pose a risk during exercise (e.g., heart conditions, severe respiratory disorders, uncontrolled hypertension).
* A history of musculoskeletal injuries or conditions that would limit participation in physical fitness activities.
* Current or recent participation in another exercise or fitness program.
* Inability to provide informed consent or unwillingness to participate voluntarily.
* Inability to provide parental consent.
* Any medical condition that contraindicates exercise or physical activity as determined by a healthcare professional.
* Age restrictions (younger than 15 and older than 18).
* Cognitive impairments that would hinder the ability to understand and follow exercise instructions.

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 77 (Actual)
Dates: Start 2024-02-10 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Affection for Physical Activity | 4 months
  Affection for Physical Activity is one of the subdomains of the Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of ten items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 50, and the minimum score is 5. The higher scores obtrained in the subdimension represent higher belief in that subscale.
Social Expectations in Physical Activity | 4 months
  Social Expectations in Physical Activity is one of the subdomains of the Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of three items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 15, and the minimum score is 3. The higher scores obtained in the subdimension represent higher belief in that subscale.
Health Expectations in Physical Activity | 4 months
  Health Expectations in Physical Activity is one of the subdomains of the Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of eight items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 40, and the minimum score is 8. The higher scores obtained in the subdimension represent higher belief in that subscale.
Attitutde towards Physical Activity | 4 months
  Attitude towards Physical Activity is a composite score of Affection for Physical Activity, Social Expectations in Physical Activity and Health Expectations in Physical Activity subdimensions of the Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of twenty-one items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 105, and the minimum score is 21. The higher scores obtained in the subdimension represent higher attitudes.
Parental Support in Physical Activity | 4 months
  Parental Support in Physical Activity is one of the subdomains of the Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of three items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 15, and the minimum score is 3. The higher scores obtained in the subdimension represent higher belief in that subscale.
Peer Support in Physical Activity | 4 months
  Peer Support in Physical Activity is one of the subdomains of Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of three items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 15, and the minimum score is 3. The higher scores obtained in the subdimension represent higher belief in that subscale.
Subjective Norms in Physical Activity | 4 months
  Subjective Norms in Physical Activity is a composite score of Parental Support in Physical Activity and Peer Support in Physical Activity, a subdimension of Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of six items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 30, and the minimum score is 6. The higher scores obtained in the subdimension represent higher attitudes.
Perceived Behavioral Control in Physical Activity | 4 months
  Perceived Behavioral Control in Physical Activity is one of the subdomains of the Physical Activity Belief Questionnaire (PAB-Q). The subscale consisted of five items answered on a 5-point Likert scale. The maximum score that can be obtained from this subscale is 25, and the minimum score is 5. The higher scores obtained in the subdimension represent higher belief in that subscale.
Body Mass Index (BMI) | 4 months
  Body Mass Index (BMI) is a numerical value derived from an individual's weight and height. The BMI is going to be expressed in units of kg/m² (kilograms per square meter) in the metric system.
Average kcals per day | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Average kilocalories (kcals) per day refer to the mean energy expenditure related to physical activity over a 24-hour period, as estimated by the wGT3X-BT accelerometer.
Time in light physical activity | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Time in light physical activity is the duration spent in activities classified as light intensity by the wGT3X-BT accelerometer.
Tme in moderate to vigorous physical activity | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Time in moderate to vigorous physical activity is the combined duration spent in activities classified as both moderate and vigorous intensity by the wGT3X-BT accelerometer.
Time in vigorous physical activity | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Time in vigorous physical activity represents the duration spent in activities classified as vigorous intensity by the wGT3X-BT accelerometer.
Time in moderate physical activity | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Time in moderate physical activity is the duration spent in activities classified as moderate intensity by the wGT3X-BT accelerometer.

SECONDARY OUTCOMES:
Body Weight | 4 months
  Body weight refers to the mass of an individual's body, and is going to measured by using Tanita BC-601 in kg.
Body Height | 4 months
  Body weight is a measurement of the vertical distance from the bottom of the feet to the top of the head when a person is standing upright. It is going to be measured by using Leicester Height Measure MK-II in m.
Activity Kilocalories | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Activity kilocalories (activity kcals), as an outcome measure from a GT3X Link accelerometer, refer to the estimated energy expenditure related to physical activity over a specified time period. The accelerometer, which records acceleration in three dimensions, allows for the assessment of different activity intensities, helping to quantify the amount of energy expended during various activities
Total Sedentary Bout | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Total sedentary bouts, as an outcome measure from a GT3X Link accelerometer, typically refer to the cumulative duration or count of extended periods of sedentary behavior detected by the accelerometer over a specified time period. Sedentary bouts are intervals during which a person is engaged in minimal or no physical activity, often characterized by activities such as sitting or lying down.
Average kcals per hour | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Average kilocalories (kcals) per hour represent the mean energy expenditure related to physical activity calculated on an hourly basis using data recorded by the wGT3X-BT accelerometer.
Total sedentary bouts | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Total sedentary bouts refer to the cumulative count or duration of extended periods of sedentary behavior detected by the wGT3X-BT accelerometer over a specified time period.
Total sedentary breaks | 4 months
  This outcome measure is going to be measured by Actigraph wGT3X-BT accelerometer. Total sedentary breaks represent the cumulative count of interruptions in sedentary behavior detected by the wGT3X-BT accelerometer over a specified time period.

CONTACTS AND LOCATIONS:
Overall Officials: Günay Yıldızer, Ph.D., Principal Investigator — Eskiehir Technical University
Locations (1):
- Eskişehir Technical University, Eskişehir, Tepebaşı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owen MB, Curry WB, Kerner C, Newson L, Fairclough SJ. The effectiveness of school-based physical activity interventions for adolescent girls: A systematic review and meta-analysis. Prev Med. 2017 Dec;105:237-249. doi: 10.1016/j.ypmed.2017.09.018. Epub 2017 Sep 28. PMID 28964852
- [Background] Belanger M, Gray-Donald K, O'Loughlin J, Paradis G, Hanley J. Influence of weather conditions and season on physical activity in adolescents. Ann Epidemiol. 2009 Mar;19(3):180-6. doi: 10.1016/j.annepidem.2008.12.008. PMID 19217000
- [Background] Kornides ML, Rimm EB, Chavarro JE, Gillman MW, Rosner B, Field AE. Seasonal Variations in Meeting Physical Activity Recommendations and Development of Overweight during Adolescence. Child Obes. 2018 Jan;14(1):33-40. doi: 10.1089/chi.2017.0118. Epub 2017 Sep 5. PMID 28872346
- [Background] Tucker P, Gilliland J. The effect of season and weather on physical activity: a systematic review. Public Health. 2007 Dec;121(12):909-22. doi: 10.1016/j.puhe.2007.04.009. Epub 2007 Oct 24. PMID 17920646
- [Background] Rowlands AV, Hughes DR. Variability of physical activity patterns by type of day and season in 8-10-year-old boys. Res Q Exerc Sport. 2006 Sep;77(3):391-5. doi: 10.1080/02701367.2006.10599373. No abstract available. PMID 17020083